CLINICAL TRIAL: NCT01645865
Title: Mobile Phone Technology for Prevention of Mother-to-Child Transmission of HIV: Acceptability, Effectiveness, and Cost
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: World Health Organization, Alliance for Health Policy and Systems Research (Unknown); Kenya National AIDS & STI Control Programme (Other)
Responsible Party: Sponsor
Other Study IDs: RPC441
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: HIV; HIV Infections; AIDS; Antiretroviral Therapy
Keywords: HIV; AIDS; PMTCT; Mobile Phone; SMS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control
  Interventions: Behavioral: Control
- Intervention
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Control — Health facilities where PMTCT services are available in the traditional clinical setting with HIV testing and counseling, PMTCT support, and enrollment in care and treatment.
  Groups: Control
Behavioral: Intervention — In addition to the 'Standard of Care', HIV-infected pregnant women and male partners within the PMTCT program are engaged in multi-directional mobile communication for PMTCT promotion with health care providers.
  Groups: Intervention

SUMMARY:
Although gains have been made in achieving the health-related Millennium Development Goals (MDG), much is still needed in countries affected by high levels of HIV/AIDS. Prevention of mother-to-child transmission (PMTCT) is a cornerstone strategy in reducing infant mortality from HIV. The study will employ a cluster randomized control trial (cRCT) with 26 health facilities randomized to two arms (intervention or control) to determine the effect of mobile phone technology on completion of key PMTCT milestones from antenatal to six weeks postpartum. The study will examine the acceptability, effectiveness, and cost of implementing a PMTCT-focused mHealth strategy among HIV-infected pregnant women, health workers, and male partners.

ELIGIBILITY:
Inclusion Criteria (female):

* HIV-positive pregnant women seeking ANC at a study site
* Up to 32 weeks gestation
* Own or have access to a mobile phone on which they can receive calls and SMS messages

Exclusion Criteria (female):

* HIV-positive pregnant women who have already initiated antiretroviral treatment

Inclusion Criteria (male):

* Referral by pregnant female partner

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants are recruited from participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The proportion of women who successfully complete key PMTCT transition points from antenatal to six weeks postpartum. | ~ 6 months
Initiation of Infant prophylaxis, Facility delivery and receipt of results of 6 weeks early infant diagnosis by DNA PCR | ~ 6 months

SECONDARY OUTCOMES:
Uptake ARV prophylaxis/ART during labor, delivery, and postpartum | ~ 6 months
Self-reported maternal adherence to ARV prophylaxis/ART during pregnancy | ~ 4 months
Time to initiation of ARV prophylaxis/ART uptake after initial identification of HIV seropositivity within ANC | ~ 1 month

CONTACTS AND LOCATIONS:
Overall Officials: John Ong'ech, MBChB, MMed, MPH, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation, UON/KNH; Seble Kassaye, MD, MS, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Elizabeth Glaser Pediatric AIDS Foundation, Nairobi, Kenya

REFERENCES:
- [Derived] Kassaye SG, Ong'ech J, Sirengo M, Kose J, Matu L, McOdida P, Simiyu R, Syengo T, Muthama D, Machekano R. Cluster-Randomized Controlled Study of SMS Text Messages for Prevention of Mother-to-Child Transmission of HIV in Rural Kenya. AIDS Res Treat. 2016;2016:1289328. doi: 10.1155/2016/1289328. Epub 2016 Dec 8. PMID 28053784